CLINICAL TRIAL: NCT03558204
Title: Surgical Management of Thumb Carpometacarpal Arthritis With Selective Joint Denervation Versus Trapeziectomy
Brief Title: Thumb Carpometacarpal Joint Denervation Versus Trapeziectomy
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00154490
Record Dates: First submitted 2018-04-05; First posted 2018-06-15 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Thumb Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CMC denervation: Patients will undergo denervation of the thumb CMC joint
  Interventions: Procedure: Denervation of the thumb CMC joint
- trapeziectomy with ligament reconstruction (LRTI): Patients will undergo excision of the trapezium and suspension of the thumb metacarpal with the flexor carpi radialis tendon
  Interventions: Procedure: trapeziectomy with ligament reconstruction (LRTI)

INTERVENTIONS:
Procedure: Denervation of the thumb CMC joint — Removal/disconnection of the nerve branches to the joint from their attachments to the joint
  Groups: CMC denervation
Procedure: trapeziectomy with ligament reconstruction (LRTI) — excision of the trapezium and suspension of the thumb metacarpal with the flexor carpi radialis tendon
  Groups: trapeziectomy with ligament reconstruction (LRTI)

SUMMARY:
This is a prospective study tracking the outcomes of patients who undergo either of two treatments for thumb carpo-metacarpal joint arthritis: trapeziectomy with ligament reconstruction (LRTI) or denervation.

DETAILED DESCRIPTION:
A total of 100 patients with carpo-metacarpal (CMC) arthritis will be enrolled in the study. The design of the study is a prospective non-blinded, non-randomized control study. Enrollment will occur at the time of initial clinic visit. All patients presenting with CMC arthritis and deemed appropriate for surgery will be considered for screened for inclusion. As a part of routine workup for CMC arthritis patients receive a hand xray. Specific attendings will perform their preferred technique for CMC arthritis: two perform denervation of the CMC joint, and two perform trapeziectomy with ligament reconstruction tendon-interposition (LRTI) only per their normal clinical practice.

Pre-operative and peri-operative care will be unchanged from standard patient care. Both procedures are outpatient procedures, usually performed under regional anesthesia and patients go home the same day. Patients are discharged with a standard thumb spica splint which is removed on their first clinic appointment which is generally post-operative day 7.

Patients enrolled in the study will have additional follow up at the 3, 6, 12 and 24 month time points. At the 3, 6, 12 and 24 month time points patients will be asked to come to clinic for evaluation with 1) a standard hand questionnaire the Michigan Hand Questionnaire, 2) lateral pinch strength, grip strength and range of motion testing, 3) Kapandji score, 4) visual analog pain scale. Each visit will take approximately 15 minutes. Patients who are unable to follow up in clinic will be given a phone questionnaire with the Michigan Hand Questionnaire, visual analog pain scale and opiate usage. There is no monetary compensation for participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women (>18 years of age) No prior traumatic thumb injuries (fractures, dislocation) No concurrent thumb procedures scheduled Eaton/Littler stage 2-4 osteoarthritis9 Minimal CMC joint subluxation on x-ray

Exclusion Criteria:

* Traumatic thumb injury (fracture, dislocation) Prior thumb surgery proximal to the interphalangeal joint. Non-fluent English Speaking Planned concurrent procedures on the thumb eg ganglion removal, trigger thumb release

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: See above
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Change in Hand Function | Through study completion at 2 years. Measurements will be performed prior to surgery, at 3 months, 6, months, 12 months, and 2 years.
  brief Michigan Hand Questionnaire (MHQ). (score ranges from 0 to 100, lower score indicates better function)
Change in grip and lateral pinch strength | Through study completion at 2 years. Measurements will be performed prior to surgery, at 3 months, 6 months, 12 months, and 2 years.
  position 2 on dynamometer (grip) and pinch meter (both are measured in kg of force, higher value indicates more strength)
Change in pain level | Through study completion at 2 years. Measurements will be performed prior to surgery, at 3 months, 6 months, 12 months, and 2 years.
  Likert scale (score ranges from 0-10, lower score indicates less pain)
narcotic pain medication usage | Up to 3 months.
  number of oxycodone 5 mg tablets (or equivalent) used after surgery (lower value indicates fewer narcotic tablets used)

SECONDARY OUTCOMES:
Time to release to unrestricted activity | Up to 6 months.
  Number of days between surgery day and when patient is released to unrestricted activity (lower value indicates fewer days between day of surgery and when the patient was released to unrestricted activity).
Operative duration | Up to 1 day
  Tourniquet time and surgery start to surgery end time (both measured in minutes, lower values indicate the surgery took less time to complete)

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Lifchez, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Haase SC, Chung KC. An evidence-based approach to treating thumb carpometacarpal joint arthritis. Plast Reconstr Surg. 2011 Feb;127(2):918-925. doi: 10.1097/PRS.0b013e3182046901. PMID 21285797
- [Result] Aliu O, Davis MM, DeMonner S, Chung KC. The influence of evidence in the surgical treatment of thumb basilar joint arthritis. Plast Reconstr Surg. 2013 Apr;131(4):816-828. doi: 10.1097/PRS.0b013e3182818d08. PMID 23542253
- [Result] Giesen T, Klein HJ, Franchi A, Medina JA, Elliot D. Thumb carpometacarpal joint denervation for primary osteoarthritis: A prospective study of 31 thumbs. Hand Surg Rehabil. 2017 Jun;36(3):192-197. doi: 10.1016/j.hansur.2017.01.007. Epub 2017 Apr 25. PMID 28465206
- [Result] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Result] Leamy DJ, Kocijan J, Domijan K, Duffin J, Roche RA, Commins S, Collins R, Ward TE. An exploration of EEG features during recovery following stroke - implications for BCI-mediated neurorehabilitation therapy. J Neuroeng Rehabil. 2014 Jan 28;11:9. doi: 10.1186/1743-0003-11-9. PMID 24468185
- [Result] Chung KC, Hamill JB, Walters MR, Hayward RA. The Michigan Hand Outcomes Questionnaire (MHQ): assessment of responsiveness to clinical change. Ann Plast Surg. 1999 Jun;42(6):619-22. doi: 10.1097/00000637-199906000-00006. PMID 10382797
- [Result] Wolf JM, Delaronde S. Current trends in nonoperative and operative treatment of trapeziometacarpal osteoarthritis: a survey of US hand surgeons. J Hand Surg Am. 2012 Jan;37(1):77-82. doi: 10.1016/j.jhsa.2011.10.010. Epub 2011 Nov 25. PMID 22119601
- [Result] Yuan F, Aliu O, Chung KC, Mahmoudi E. Evidence-Based Practice in the Surgical Treatment of Thumb Carpometacarpal Joint Arthritis. J Hand Surg Am. 2017 Feb;42(2):104-112.e1. doi: 10.1016/j.jhsa.2016.11.029. PMID 28160900
- [Result] Waljee JF, Chung KC. Outcomes research in rheumatoid arthritis. Hand Clin. 2011 Feb;27(1):115-26. doi: 10.1016/j.hcl.2010.10.005. PMID 21176806